CLINICAL TRIAL: NCT01666548
Title: Haemolytic Uraemic Syndrome in Childhood: Clinical, Cognitive and Psychological Aspects
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2011-0394
Record Dates: First submitted 2012-07-31; First posted 2012-08-16 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Hemolytic-Uremic Syndrome; Children; Parents; Psychological Adjustment
Keywords: haemolytic uraemic syndrome; complications of HUS; renal replacement treatment; renal function outcome; neuropsychological sequelae; psychological adjustment; quality of life
MeSH Terms: conditions — Hemolytic-Uremic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — urine, native-blood, blood plasma, EDTA stabilized blood, heparin blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the clinical, cognitive outcome and psychosocial outcome of haemolytic uraemic syndrome in childhood.

The haemolytic uraemic syndrome (HUS) is the leading cause of acute renal failure in childhood. The more common typical HUS is mostly caused by Shigatoxin-producing enterohaemorrhagic Escherichia coli (EHEC). The rarer atypical HUS is mainly caused by different genetic abnormalities in complement regulatory proteins.

About 50 till 60 percent of all patients with HUS develop a severe acute renal failure and require dialysis. Resulting from new diagnostic and therapeutic approaches the survival rate increased during the last years. Despite this, there are only few data concerning long-term prognosis, cognitive and motoric development, as well as psychological coping and health-related quality of life of affected children and their parents.

DETAILED DESCRIPTION:
The main purposes of this study are: the evaluation of the long-term renal function of pediatric HUS-patients; the evaluation of the dialysis method in the acute phase of the disease and its impact on the duration of the renal-placement-therapy, as well as the long-term renal function; the evaluation of the intellectual and motoric performance of affected children and the evaluation of the health-related quality of life and psychological processing of the patients themselves and their parents.

All cases of HUS treated at the University Children's Hospital Zurich between 1995 and 2012 will be analyzed retrospectively. In the course of a routine-follow-up-examination the clinical data of patients up to the age of 17 years will be actualized and completed. The results of clinical and paraclinical investigations related to renal function will be evaluated to describe the clinical features of haemolytic uraemic syndrome in childhood.

Intellectual performance will be analyzed with the Wechsler-Intelligence Scale for Children-IV (WISC-IV) and motoric performance with the Zurich Neuromotor Assessment in children at the age from 6 to 16 years.

The health-related quality-of-life of all parents and affected children from the age of 7 years will be assessed by different generic quality-of-life-instruments.

ELIGIBILITY:
Inclusion Criteria:

* children and youth from 2 months to 17 years who had suffered from haemolytic uraemic syndrome
* willingness and ability to participate in the study
* freely signed informed consent

Exclusion Criteria:

* missing written informed consent
* children who do not fulfil the age criterion

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children and youth from 2 months to 17 years in who had suffered from haemolytic uraemic syndrome
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
- renal function (estimated glomerular filtration rate according to the SCHWARTZ formula) after haemolytic uraemic syndrome in childhood | 1 year 5 months
- quality of life of children with haemolytic uraemic syndrome and their parents | 1 year 5 months
- neuropsychological sequelae of children with haemolytic uraemic syndrome | 1 year 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Spartà, MD, Principal Investigator — Nephrology Unit, University Children's Hospital, Zurich, Steinwiesstrasse 75, CH-8032 Zürich, Switzerland
Locations (1):
- Nephrology Unit of the University Children's Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Neuhaus TJ, Calonder S, Leumann EP. Heterogeneity of atypical haemolytic uraemic syndromes. Arch Dis Child. 1997 Jun;76(6):518-21. doi: 10.1136/adc.76.6.518. PMID 9245850
- [Background] Brunner K, Bianchetti MG, Neuhaus TJ. Recovery of renal function after long-term dialysis in hemolytic uremic syndrome. Pediatr Nephrol. 2004 Feb;19(2):229-31. doi: 10.1007/s00467-003-1337-4. Epub 2003 Nov 27. PMID 14648326
- [Background] Ruth EM, Landolt MA, Neuhaus TJ, Kemper MJ. Health-related quality of life and psychosocial adjustment in steroid-sensitive nephrotic syndrome. J Pediatr. 2004 Dec;145(6):778-83. doi: 10.1016/j.jpeds.2004.08.022. PMID 15580200
- [Background] Falger J, Latal B, Landolt MA, Lehmann P, Neuhaus TJ, Laube GF. Outcome after renal transplantation. Part I: intellectual and motor performance. Pediatr Nephrol. 2008 Aug;23(8):1339-45. doi: 10.1007/s00467-008-0795-0. Epub 2008 Apr 4. PMID 18389283
- [Background] Falger J, Landolt MA, Latal B, Ruth EM, Neuhaus TJ, Laube GF. Outcome after renal transplantation. Part II: quality of life and psychosocial adjustment. Pediatr Nephrol. 2008 Aug;23(8):1347-54. doi: 10.1007/s00467-008-0798-x. Epub 2008 Apr 3. PMID 18386069
- [Background] Schifferli A, von Vigier RO, Fontana M, Sparta G, Schmid H, Bianchetti MG, Rudin C; Swiss Pediatric Surveillance Unit. Hemolytic-uremic syndrome in Switzerland: a nationwide surveillance 1997-2003. Eur J Pediatr. 2010 May;169(5):591-8. doi: 10.1007/s00431-009-1079-9. Epub 2009 Oct 15. PMID 19830454
- [Background] Pollock KG, Duncan E, Cowden JM. Emotional and behavioral changes in parents of children affected by hemolytic-uremic syndrome associated with verocytotoxin-producing Escherichia coli: a qualitative analysis. Psychosomatics. 2009 May-Jun;50(3):263-9. doi: 10.1176/appi.psy.50.3.263. PMID 19567766
- [Background] Schlieper A, Orrbine E, Wells GA, Clulow M, McLaine PN, Rowe PC. Neuropsychological sequelae of haemolytic uraemic syndrome. Investigators of the HUS Cognitive Study. Arch Dis Child. 1999 Mar;80(3):214-20. doi: 10.1136/adc.80.3.214. PMID 10325699
- [Derived] Buder K, Werner H, Landolt MA, Neuhaus TJ, Laube GF, Sparta G. Health-related quality of life and mental health in parents of children with hemolytic uremic syndrome. Pediatr Nephrol. 2016 Jun;31(6):923-32. doi: 10.1007/s00467-015-3294-0. Epub 2015 Dec 23. PMID 26701835